CLINICAL TRIAL: NCT03253991
Title: A Study to Evaluate the Effectiveness and Safety of ExAblate Transcranial MRgFUS Thalamotomy Treatment of Medication Refractory Essential Tremor Subjects
Brief Title: A Study to Evaluate the Effectiveness and Safety of ExAblate MRgFUS on Essential Tremor
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET002J
Record Dates: First submitted 2017-07-24; First posted 2017-08-18 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Intervention Model Description: Prospective multi-site, single-arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRgFUS treatment (Experimental): MRgFUS device treatment, thalamotomy
  Interventions: Device: MRgFUS treatment

INTERVENTIONS:
Device: MRgFUS treatment — ExAblate Transcranial MRgFUS Thalamotomy Treatment of Medication Refractory Essential Tremor Subjects
  Other Names: Thalamotomy

SUMMARY:
A Study to Evaluate the Effectiveness and Safety of ExAblate Transcranial MRgFUS Thalamotomy Treatment of Medication Refractory Essential Tremor Subjects

The objective of this prospective, single-arm study is to test the efficacy of treatment using the ExAblate Transcranial System and to further demonstrate safety in medication-refractory tremor inpatients with essential tremor (ET).

The Indications for Use claim for this system is as follows: Treatment of medication-refractory tremor in patients with essential tremor.

DETAILED DESCRIPTION:
The objective of this prospective, multi-site, single-arm study is to test the efficacy of treatment using the ExAblate Transcranial System and to further demonstrate safety in medication-refractory tremor in subjects with essential tremor (ET).

Safety: To evaluate the incidence and severity of adverse events (AE/AEs) associated with ExAblate Transcranial MRgFUS treatment of medication-refractory ET Effectiveness: To determine the effectiveness of the ExAblate Transcranial MRgFUS treatment of medication-refractory tremor (i.e. ET). Efficacy will be determined utilizing the Clinical Rating Scale for Tremor (CRST) in ET from examinations at baseline and 3-Months post-ExAblate treatment.

• This study is designed as a prospective, multi-site, single-arm study. Assessments of primary efficacy endpoints will compare the three months after ExAblate treatment to Baseline measurements for clinical symptom relief. Safety of ExAblate in the treatment of ET will be collected for one year after ExAblate treatment. Relative Safety will be evaluated using a common description of Significant Clinical Complications for patients treated in this study. This study will be performed on the 3T MR scanners.

The secondary endpoints of the study are as follows:

1. Quality life claims: Questionnaire for Essential Tremor (QUEST) outcome (upper extremity questions) at Months 3 change from Baseline
2. Durability (as measured by QUEST upper arm extremity questions) of the procedure as reflected by the efficacy data through change from baseline measures through Month 12 follow up
3. Subject daily functionalities: as measured by CRST Part-C (subscales)Month 12 as compared to Baseline.

ELIGIBILITY:
Inclusion Criteria

* Men and women age 22 years or older
* A diagnosis of ET as confirmed from clinical history and examination by a neurologist or neurosurgeon specialized in movement disorder
* Have had an inadequate response to one or two oral doses of medication, per local standards. An inadequate medication trial is defined as a therapeutic dose of each medication and poor response to drug, or the development of side effects as the medication dose is titrated.
* Able to communicate sensations during the ExAblate TcMRgFUS treatment

Exclusion criteria:

* Subjects with unstable cardiac status
* Severe hypertension (diastolic BP > 100 on medication)
* Subjects with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
* Known intolerance or allergies to the MRI contrast agent (e.g. Gadolinium or Magnevist) including advanced kidney disease
* Patient with severely impaired renal function
* History of abnormal bleeding and/or coagulopathy
* History of immunocompromise including those who are HIV positive.
* History of intracranial hemorrhage
* Cerebrovascular disease (multiple CVA or CVA within 6 months)
* Subjects with uncontrolled symptoms and signs of increased intracranial pressure (e.g., headache, nausea, vomiting, lethargy, papilledema).
* Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment (can be up to 4 hrs of total table time.)
* Are participating or have participated in another clinical trial in the last 30 days
* Significant claustrophobia that cannot be managed with mild medication.
* Presence of any other neurodegenerative disease such as Parkinson-plus syndromes suspected on neurological examination.
* Presence of significant cognitive impairment
* Subjects with life-threatening systemic disease
* Subjects with a history of seizures within the past year
* Subjects with presence or history of psychosis

Ages: 22 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2014-11-17 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Safety - Will be determined evaluating incidence and severity of device related complications from first treatment day visit through all follow ups. Relative Safety will be evaluated describing Significant Clinical Complications for patients treated. | 1 year
  All AEs will be reported and categorized by investigators as definitely, probably, possibly, or unrelated to the device or procedure and categorized by treatment group / treatment arm. Relative Safety will be evaluated using a common description of Significant Clinical Complications for patients treated in this study.
Effectiveness - Will be evaluated using the Clinical Rating Scale for Tremors (CRST) for ET subjects. Comparison will be performed from examinations at baseline and 3-Months post-ExAblate treatment. | 5 Years
  Assessments of efficacy endpoints will compare the three months after ExAblate treatment to Baseline measurements for clinical symptom relief.

CONTACTS AND LOCATIONS:
Locations (11):
- China (2):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Henan Provincial People's Hospital, Zhengzhou, Henan
- Japan (8):
  - Sadamoto Hospital, Ehime
  - Shonan Fujisawa Tokushukai Hospital, Fujisawa
  - Hokkaido Ohno Memorial Hospital, Hokkaido
  - Hokuto, Hokkaido
  - Ohanishi Noerological Center, Hyōgo
  - Kumagaya General Hospital, Kumagaya
  - Department of Neurosurgery, Osaka University Hospital, Osaka
  - Tokyo Women's Medical University Hospital, Tokyo
- Chang Bing Show Chwan Memorial Hospital, Chang-hua, Taiwan

REFERENCES:
- [Derived] Zong R, Li X, Yin C, He J, Zhang D, Bian X, Huang L, Zhou J, Ling Z, Ma L, Lou X, Pan L, Yu X. Magnetic resonance-guided focused ultrasound for essential tremor: a prospective, single center, single-arm study. Neural Regen Res. 2024 Sep 1;19(9):2075-2080. doi: 10.4103/1673-5374.391192. Epub 2024 Jan 12. PMID 38227538